CLINICAL TRIAL: NCT01888575
Title: Assessment of Low-dose ASA Discontinuation Risk Associated With Concomitant PPI Use During the First Year of ASA Therapy for Secondary Prevention
Brief Title: Assessment of Low-dose ASA Discontinuation Risk Associated With Concomitant PPI Use During the First Year of ASA Therapy
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5040N00008
Record Dates: First submitted 2013-03-18; First posted 2013-06-28 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Cardiovascular Prevention
Keywords: Discontinuation of low dose ASA,; Secondary cardiovascular prevention,; Acid-suppressing drugs,; Gastrointestinal risk,; Epidemiology
MeSH Terms: interventions — Risk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Aspirin discontinuers; Aspirin non-discontinuers: Patients on low dose ASA for secondary prevention that discontinue aspirin and those not discontinuing aspirin
  Interventions: Drug: Risk of low dose aspirin discontinuation
- Drug: PPI continuous use; No PPI use

INTERVENTIONS:
Drug: Risk of low dose aspirin discontinuation — PPI continuous use; No PPI usePPI
  Groups: Aspirin discontinuers; Aspirin non-discontinuers

SUMMARY:
This study is conducted in a cohort of low dose aspirin (ASA) users previously ascertained .The aims of the post hoc analyses are:

To estimate the one year risk of discontinuation of use of low-dose ASA associated to PPI concomitant use versus non-use, crude and adjusted by confounding.

To estimate the one year risk of discontinuation of use of low-dose ASA associated to PPI concomitant use stratified by age and sex.

To evaluate other predictors of discontinuation of low-dose ASA during the first year of ASA therapy.

DETAILED DESCRIPTION:
Assessment of low-dose ASA discontinuation risk associated with concomitant PPI use during the first year of ASA therapy for secondary prevention

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50-84 years in 2000-2007.
* Patients with first prescription of low dose ASA ( see study population description).
* Patients were required to have been enrolled with their primary care practitioner (PCP) for at least 2 years and to have a computerized prescription history of at least 1 year before the start of the study.

Exclusion Criteria:

* Patients aged below age 50 and 85 years and above ( see study population description).
* Patients with a diagnosis of cancer, alcohol abuse or alcohol-related disease.
* Incomplete data recording in THIN.

Ages: 50 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a pharmacoepidemiology study using data from The Health Improvement Network (THIN) primary care database in the UK. Patients aged 50-84 years with evidence of ischemic heart disease or cerebrovascular disease, who were new users of low-dose ASA (75-300 mg/day) and who had received at least two low-dose ASA prescriptions for the secondary prevention of cardiovascular disease or cerebrovascular disease between 2000 and 2007 were identified from THIN. .
Sampling Method: Non-Probability Sample
Enrollment: 35604 (Actual)
Dates: Start 2012-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Risk of low dose ASA discontinuation associated with continuous PPI use vs.non-use | Up to 1 year.
  Risk (hazard ratios) of low dose ASA discontinuation associated with continuous PPI use vs. non-use.
Risk of low dose ASA discontinuation associated with baseline gastrointestinal risk category ( high risk versus low risk) | Up to 1 year
  Risk ( hazard ratios) of low dose ASA discontinuation associated with baseline gastrointestinal risk category( high risk versus low risk).

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Garcia Rodriguez, MD, Principal Investigator — CEIFE (Centro Espanol de Investigacion Farmacoepidemiologica - Spanish Centre for Pharmacoepidemiologic Research )
Locations (1):
- Research Site, Madrid, Spain

REFERENCES:
- [Background] Cea Soriano L, Rodriguez LA. Risk of Upper Gastrointestinal Bleeding in a Cohort of New Users of Low-Dose ASA for Secondary Prevention of Cardiovascular Outcomes. Front Pharmacol. 2010 Oct 14;1:126. doi: 10.3389/fphar.2010.00126. eCollection 2010. PMID 21811460
- [Background] Garcia Rodriguez LA, Cea Soriano L, Hill C, Johansson S. Increased risk of stroke after discontinuation of acetylsalicylic acid: a UK primary care study. Neurology. 2011 Feb 22;76(8):740-6. doi: 10.1212/WNL.0b013e31820d62b5. Epub 2011 Jan 26. PMID 21270415
- See also: D5040N00008_CSP.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=463&filename=D5040N00008_CSP.pdf